CLINICAL TRIAL: NCT00933751
Title: Changes of Oxygen Saturation in Inferior Vena Cava (IVC) in Patients During and After High Risk Abdominal Surgery and Relationship to the Outcome.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Changes of the oxygen saturation in the IVC during and after major abdominal surgery and relationship to the outcome, Zoya Haitov MD
Other Study IDs: 100/09
Record Dates: First submitted 2009-07-05; First posted 2009-07-07 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2009-07

CONDITIONS: Abdominal Surgery
Keywords: central venous oxygen saturation; oxygen transport; physiologic monitoring; tissue oxygenation; Patients before high risk abdominal surgery
MeSH Terms: interventions — Catheterization, Central Venous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients before emergent major abdominal surgery
  Interventions: Device: Central vein catheterization

INTERVENTIONS:
Device: Central vein catheterization — Blood samplings from IVC catheter

SUMMARY:
Tissue hypoxia is one of the most important factors leading to the development of multiorgan failure. Patients presenting for emergent major abdominal surgery might suffer from organ hypoperfusion. Thus, early detection of the imbalance between oxygen supply and demand may improve the outcome. The investigators believe that hypoperfusion of the abdominal organs will cause a decrease of the saturation in the hepatic vein and in the IVC.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients presenting for emergency surgery due to acute abdomen pain
* Older than 18 years old
* Not pregnant

Exclusion Criteria:

* Age < 18
* Pregnancy
* Major coagulopathy
* Permanent pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients before emergent high risk abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh MC, Beer-Yaakov, Israel